CLINICAL TRIAL: NCT05158738
Title: Inherited Cardiac cONditions In Kids: Understanding the Genetics and Outcomes of Paediatric Inherited CardiacConditions
Brief Title: Inherited Cardiac cONditions In Kids
Acronym: ICONIK
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 288514
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Inherited Cardiac Conditions; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Age of Onset

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — 1. Blood- plasma and serum
  2. Saliva
  3. Collection of additional tissue samples (myocardial, skeletal, skin) from planned clinical procedures (where applicable)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients with inherited cardiac condition, onset <16 years old and Parents — Patients with a confirmed diagnosis of an inherited cardiac condition, onset <16 years old and Parents will have samples that undergo whole genome sequencing and biomarker analysis

SUMMARY:
All patients with heart disease should have the opportunity to participate in research into their condition, to advance knowledge and treatment. The investigators have built an online registry and database - The Heart Hive - to connect research-willing participants (with heart muscle disease) with active researchers and projects. Participants enrol and upload their own data through the website.This study uses The Heart Hive platform to study cardiomyopathies - heart muscle disease. These are progressive diseases, and there is a need to better understand what factors affect the chances of developing cardiomyopathy, and how the condition progresses. The study will collect information about participants diagnosis, DNA for genetic analysis, and then follow participants' clinical progress. The study will identify genetic variants that cause cardiomyopathy, and determine which specific genetic or environmental factors predict disease severity, progression and response to treatment, with an overall objective of identifying new and personalised treatments for patients with this disease.

DETAILED DESCRIPTION:
This is a multi-centre, observational study of children with rare inherited cardiac conditions. The focus of the study will be on children with clinically diagnosed cardiomyopathy and their unaffected parents, with collection of baseline demographic data, imaging data, and genotyping data. Children and their parents will been rolled over a 5-year period.

Sub-sets of patients with confirmed diagnoses of other heritable cardiovascular diseases with onset <16 years will also be recruited.These will include children who following evaluation by their clinical multidisciplinary team (which will include a geneticist or genetic counsellor) are likely to have a rare monogenic condition. Other affected family members of eligible patients may be also invited to participate in the study.

Information for this study will be collected primarily from investigations performed as part of the participants' routine clinical care including whole genome sequencing commissioned by NHS England. The study will seek consent to access and export this data. Procedures performed as part of this study may include venepuncture and/or saliva collection and carry minimal risk to the patient.

Parents of participants that are recruited into the study will donate a blood sample (or saliva sample if unable to provide blood) and consent will be requested for collection of health information and results of relevant investigations carried out as part of their routine clinical care (e.g. an echocardiogram). Other family members that are recruited into the study will donate a blood sample (or saliva sample if unable to provide blood) and consent will be requested for collection of health information. Family members of deceased patients with cardiomyopathy or other inherited cardiac conditions may be asked if they wish to donate stored samples that may have been taken prior to death or as part of a post-mortem examination to establish cause of death. Any discussion with regard to the use of stored samples for this project will be initiated by the clinical care team for the deceased patient and their family to minimise any potential distress to the family. Sub-sets of patients may be asked to donate tissue samples taken as part of their clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with a confirmed diagnosis of childhood onset (<16 years) PCM
* Males or females with childhood onset (<16 years) of a rare inherited cardiac condition likely to be a monogenic condition
* Capacity for parents to provide informed consent
* Genotype negative following local standard diagnostic ICC gene panel
* Family members of patients with ICC, both affected and unaffected

Exclusion Criteria:

* Parents who lack capacity to provide consent on behalf of their children/themselves
* Onset over 16 years
* Significant teratogen exposure (including maternal diabetes) likely to contribute to cardiac dysfunction (following discussion with Cardiologist)
* Significant coronary heart disease likely to contribute to cardiac dysfunction (following discussion with Cardiologist)
* Other secondary causes of cardiac dysfunction likely to explain the phenotype of the patient
* Patients with a confirmed genetic diagnosis (patients with variants of uncertain significance are not excluded).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Males or females with a confirmed diagnosis of childhood onset (<16 years) PCM and their parents.
  * Males or females with childhood onset (<16 years) of a rare inherited cardiac condition likely to be a monogenic condition and their parents.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measures | 5 years
  Identification of novel genetic variants associated with disease status or outcome

CONTACTS AND LOCATIONS:
Overall Officials: James Ware, Principal Investigator — Imperial College London
Locations (3):
- United Kingdom (3):
  - Royal Brompton Hospital, London
  - Great Ormond Street Hospital for Children, London
  - Harefield Hospital, Uxbridge

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries will be shared with collaborating sites
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: During planning (December 2021) and throughout the study recruitment and follow-up period
Access Criteria: Provided through secure data transfer mechanisms approved by Imperial College London and secure email